CLINICAL TRIAL: NCT05599945
Title: A First Human Dose Study Investigating Safety, Tolerability, and Pharmacokinetics of Single Subcutaneous Injections of NNC0581-0001 in Healthy Adults and in Participants With Hepatic Steatosis
Brief Title: First Human Dose Trial for a New Medication to Potentially Treat Liver Diseases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN6581-4860; U1111-1274-4577 (Other: World Health Organization (WHO)); 2022-001359-18 (EudraCT Number)
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Healthy Volunteers; Hepatic Steatosis
MeSH Terms: conditions — Fatty Liver

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Single Dose 1: NNC0581-0001 10 milligram (mg) (Experimental): Part A: Healthy participants will receive a single dose of NNC0581-0001 10 mg or matching placebo injection subcutaneously.
  Interventions: Drug: NNC0581-0001; Drug: Placebo (NNC0581-0001)
- Single Dose 2: NNC0581-0001 30 mg (Experimental): Part A: Healthy participants will receive a single dose of NNC0581-0001 30 mg or matching placebo injection subcutaneously.
  Interventions: Drug: NNC0581-0001; Drug: Placebo (NNC0581-0001)
- Single Dose 3: NNC0581-0001 90 mg (Experimental): Part A: Healthy participants will receive a single dose of NNC0581-0001 90 mg or matching placebo injection subcutaneously.
  Interventions: Drug: NNC0581-0001; Drug: Placebo (NNC0581-0001)
- Single Dose 4: NNC0581-0001 250 mg (Experimental): Part A: Healthy participants will receive a single dose of NNC0581-0001 250 mg or matching placebo injection subcutaneously.
  Interventions: Drug: NNC0581-0001; Drug: Placebo (NNC0581-0001)
- Single Dose 5: NNC0581-001 600 mg (Experimental): Part B: Participants with hepatic steatosis will receive a single dose of NNC0581-0001 600 mg or matching placebo injection subcutaneously.
  Interventions: Drug: NNC0581-0001; Drug: Placebo (NNC0581-0001)
- Single Dose 6: NNC0581-001 1000 mg (Experimental): Part B: Participants with hepatic steatosis will receive a single dose of NNC0581-0001 1000 mg or matching placebo injection subcutaneously.
  Interventions: Drug: NNC0581-0001; Drug: Placebo (NNC0581-0001)

INTERVENTIONS:
Drug: NNC0581-0001 — Participants will receive up to six single dose levels of subcutaneous NNC0581-0001 in a sequential manner with the dose increasing between cohorts.
Drug: Placebo (NNC0581-0001) — Participants will receive single dose of subcutaneous injection of placebo matched to NNC0581-0001.

SUMMARY:
This study will assess the safety, tolerability, the pharmacokinetics from single injection (under the skin) of NNC0581-0001 and explores the pharmacodynamics in healthy participants and participants with hepatic steatosis (increased liver fat). Participants will either get NNC0581-001 or Placebo (dummy treatment). Which treatment participants get is decided by chance.NNC0581-0001 is a new medicine which cannot be prescribed by doctors. The study will last about 58 weeks.

ELIGIBILITY:
Inclusion Criteria, for healthy participants in Part A:

* Female of non-childbearing potential or male aged 18-55 years (both inclusive) at the time of signing informed consent.
* Body Mass Index (BMI) from 18.5 to 30.0 kilogram per square meter (kg/m^2) (both inclusive) at screening.
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram, and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Inclusion criteria for participants with hepatic steatosis in Part B:

* Female of non-childbearing potential or male aged 18-55 years (both inclusive) at the time of signing informed consent.
* Body Mass Index (BMI) from 25.0 to 34.9 kilogram per square meter (kg/m^2) (both inclusive) at screening.
* Hepatic steatosis identified by a score above 248 dB/m by Fibroscan® (Controlled Attenuated Parameter, CAP) at screening.

Exclusion Criteria

* Any disorder, which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol.
* For Part A: Any laboratory safety parameters at screening outside the below laboratory ranges, see laboratory provided reference ranges for specific values (re-screening or re-sampling is NOT allowed if the participant has failed one of the exclusion criteria related to laboratory parameters):
* Alanine aminotransferase (ALT) greater than upper normal limit (UNL) plus 10 percent
* Aspartate aminotransferase (AST) greater than UNL plus 10 percent
* Bilirubin greater than UNL plus 10 percent
* Estimated glomerular filtration rate (eGFR) below 90 milliliters per minute per 1.73 square meters (90 mL/min/1.73m^2)
* Glycated haemoglobin (HbA1c) greater than or equal to 5.7 percent (39 millimole per mole [mmol/mol]) at screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2022-11-23 (Actual); Primary Completion 2025-08-29 (Actual); Study Completion 2025-08-29 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAEs) | From dosing (Day 1) until completion of the End of Study Visit at week 52
  Measured as number of events.

SECONDARY OUTCOMES:
AUC0-∞: The area under the NNC0581-0001 plasma concentration-time curve from time zero to infinity after a single dose | From dosing (Day 1) to 168 hours after dosing
  Measured in nanogram hour per mililiter (ng*h/mL).
Cmax: The maximum concentration of NNC0581-0001 in plasma after a single dose | From dosing (Day 1) to 168 hours after dosing
  Measured in nanogram per mililiter (ng/mL).
tmax: The time from dose administration to maximum plasma concentration of NNC0581-0001 after a single dose | From dosing (Day 1) to 168 hours after dosing
  Measured in Hours.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (2):
- United Kingdom (2):
  - Parexel CPRU, Level 7, Harrow, Middlesex
  - Parexel Research Unit, Harrow, Middlesex

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com.